CLINICAL TRIAL: NCT01412801
Title: A Phase II Open-Label, Multi-Center Study of a Group B Streptococcus Vaccine in HIV Positive and HIV Negative Pregnant Women
Brief Title: Magnitude of the Antibody Response to and Safety of a GBS Trivalent Vaccine in HIV Positive and HIV Negative Pregnant Women and Their Offsprings
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V98_05
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Streptococcal Infections; Gram-Positive Bacterial Infections; Bacterial Infections
Keywords: Group B streptococcus; GBS; Vaccine; Prevention of group B streptococcus infection
MeSH Terms: conditions — Streptococcal Infections; Gram-Positive Bacterial Infections; Bacterial Infections

ARMS (3):
- HIVneg (Experimental): HIV-antibody negative maternal subjects at 24 to 35 weeks gestation received one dose of Group B streptococcus vaccine.
  Interventions: Biological: Group B streptococcus vaccine
- HIVposCD4HIGH (Experimental): HIV-antibody positive maternal subjects at 24 to 35 weeks gestation with CD4+ count >350 cells/µL received one dose of Group B streptococcus vaccine.
  Interventions: Biological: Group B streptococcus vaccine
- HIVposCD4LOW (Experimental): HIV-antibody positive maternal subjects at 24 to 35 weeks gestation with CD4+ count ≤350 cells/µL but > 50 cells/µL received one dose of Group B streptococcus vaccine
  Interventions: Biological: Group B streptococcus vaccine

INTERVENTIONS:
Biological: Group B streptococcus vaccine — Subjects receive one dose of 5 μg of each of the 3 glycoconjugates present in the Group B streptococcus vaccine.

SUMMARY:
The study compared the magnitude of the antibody response and safety of a GBS Trivalent Vaccine in HIV positive and HIV negative pregnant women and their offspring. In addition the study investigated the maternal to fetal transfer of antibodies induced by the investigational vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18-40 years of age between 24-35 weeks gestation
* Women who were HIVneg or HIVpos with WHO stage I or II disease and with CD4+ counts > 50 cells/µL

Exclusion Criteria:

* Women who had CD4+ count ≤ 50 cells/µL
* Women who were HIVpos with WHO stage III or IV disease, history of severe allergic reactions after previous vaccinations

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (2):
- Limbe Health Center, Blantyre, Malawi
- Chris Hani Baragwanath Hospital, Bertsham, South Africa

REFERENCES:
- [Derived] Heyderman RS, Madhi SA, French N, Cutland C, Ngwira B, Kayambo D, Mboizi R, Koen A, Jose L, Olugbosi M, Wittke F, Slobod K, Dull PM. Group B streptococcus vaccination in pregnant women with or without HIV in Africa: a non-randomised phase 2, open-label, multicentre trial. Lancet Infect Dis. 2016 May;16(5):546-555. doi: 10.1016/S1473-3099(15)00484-3. Epub 2016 Feb 8. PMID 26869376

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at Malawi and South Africa
Pre-assignment Details: All the enrolled subjects are included in the trial. Also,only the mothers who received the glycoconjugates were considered enrolled.
Groups:
- HIVposCD4LOW_Maternal: HIV-antibody positive maternal subjects at 24 to 35 weeks gestation with CD4+ count ≤350 cells/µL but > 50 cells/µL received one dose of 5 μg of each of the 3 glycoconjugates present in the GBS Trivalent Vaccine
- HIVposCD4HIGH_Maternal: HIV-antibody positive maternal subjects at 24 to 35 weeks gestation with CD4+ count >350 cells/µL received one dose of 5 μg of each of the 3 glycoconjugates present in the GBS Trivalent Vaccine
- HIVneg_Maternal: HIV-antibody negative maternal subjects at 24 to 35 weeks gestation received one dose of 5 μg of each of the 3 glycoconjugates present in the GBS Trivalent Vaccine
- HIVposCD4LOW(Infants): Infants born to HIV-antibody positive maternal subjects with CD4+ count ≤350 cells/µL but > 50 cells/µL .
- HIVposCD4HIGH(Infants): Infants born to HIV-antibody positive maternal subjects with CD4+ count >350 cells/µL
- HIVneg(Infants): Infants born to HIV-antibody negative maternal subjects
Period: Overall Study
Arm/Group | HIVposCD4LOW_Maternal | HIVposCD4HIGH_Maternal | HIVneg_Maternal | HIVposCD4LOW(Infants) | HIVposCD4HIGH(Infants) | HIVneg(Infants)
Started | 91 | 89 | 90 | 91 | 88 | 87
Completed | 87 | 84 | 83 | 87 | 85 | 84
Not Completed | 4 | 5 | 7 | 4 | 3 | 3
Not completed — Death | 0 | 1 | 0 | 4 | 2 | 2
Not completed — Lost to Follow-up | 1 | 2 | 4 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 1 | 0 | 0 | 0
Not completed — Relocated to another area | 0 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- HIVposCD4LOW (Infants): Infants born to HIV-antibody positive maternal subjects with CD4+ count ≤350 cells/µL but > 50 cells/µL
- HIVposCD4HIGH (Infants): Infants born to HIV-antibody positive maternal subjects with CD4+ count >350 cells/µL
- HIVneg (Infants): Infants born to HIV-antibody negative maternal subjects
- Total: Total of all reporting groups
Arm/Group | HIVposCD4LOW_Maternal | HIVposCD4HIGH_Maternal | HIVneg_Maternal | HIVposCD4LOW (Infants) | HIVposCD4HIGH (Infants) | HIVneg (Infants) | Total
Number analyzed (Participants) | 91 | 89 | 90 | 91 | 88 | 87 | 536
Age, Customized [Mean (Standard Deviation); unit: years]
  Maternal Subjects | 28.3 (4.8) | 28.1 (5.2) | 24.7 (4.4) | NA (NA) — "Mothers' ages only provided Here" | NA (NA) — "Mothers' ages only provided Here" | NA (NA) — "Mothers' ages only provided Here" | 27.1 (5.0)
Age, Customized [Mean (Standard Deviation); unit: days]
  Infants | NA (NA) — "Infants' ages only provided here" | NA (NA) — "Infants' ages only provided here" | NA (NA) — "Infants' ages only provided here" | 4.1 (1.6) | 6.7 (2.5) | 1.3 (1.1) | 1.6 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 89 | 90 | 42 | 40 | 41 | 393
  Male | 0 | 0 | 0 | 49 | 48 | 46 | 143

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentrations (GMCs) of Antibodies in Maternal Subjects and Infants at Delivery/Birth
Description: GMCs of Group B Streptococcus (GBS)-specific Abs against serotypes Ia, Ib and III in mothers and in infants at delivery/birth are presented.
Time Frame: Day of delivery/birth
Population: Full Analysis Set (FAS)-Maternal and Infant Subjects: Maternal subjects provided at least one evaluable serum sample result at delivery; infant subjects provided at least one evaluable sample result at birth (from cord blood, or peripheral blood within 72 hours when cord blood was unavailable).
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | HIVposCD4LOW_Maternal | HIVposCD4HIGH_Maternal | HIVneg_Maternal | HIVposCD4LOW(Infants) | HIVposCD4HIGH(Infants) | HIVneg(Infants)
Number analyzed (Participants) | 83 | 81 | 83 | 83 | 81 | 83
μg/mL
  GBS serotypes Ia (83, 81, 83, 79, 81, 83) | 2.07 [1.44 to 2.98] | 2.31 [1.6 to 3.34] | 3.98 [2.75 to 5.74] | 1.01 [0.66 to 1.56] | 1.22 [0.8 to 1.87] | 3.91 [2.56 to 5.96]
  GBS serotypes Ib(74, 80, 82, 44, 56, 57) | 1.84 [1.22 to 2.77] | 2.4 [1.64 to 3.52] | 4.08 [2.85 to 5.83] | 1.31 [0.78 to 2.19] | 1.62 [1.03 to 2.56] | 2.67 [1.7 to 4.2]
  GBS serotypes III (83, 72, 82, 54, 51, 66) | 1.07 [0.71 to 1.6] | 1.03 [0.69 to 1.53] | 3.61 [2.51 to 5.18] | 0.6 [0.36 to 0.99] | 0.52 [0.31 to 0.88] | 3.88 [2.47 to 6.1]

2. Secondary Outcome: Vaccine Induced Maternal Serotype Specific GBS Antibody Levels for GBS Serotypes Ia, Ib and III at Day 1, 15, 31 and at Delivery
Description: Immunogenicity was measured as Geometric Mean Concentration of Antibody levels for GBS Serotypes Ia, Ib and III after receiving one dose of GBS Trivalent Vaccine.
Time Frame: Day 1, 15, 31 and at Delivery
Population: FAS (Maternal Subjects in the Exposed Population) who -Secondary objective serum GMC: provided at least one evaluable sample result at day 1 (prior to vaccination), day 15, day 31, or at delivery;- Secondary objective kinetics: provided at least one evaluable serum sample at day 1 (prior to vaccination), day 15, day 31, and at delivery.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | HIVposCD4LOW_Maternal | HIVposCD4HIGH_Maternal | HIVneg_Maternal
Number analyzed (Participants) | 74 | 75 | 77
µg/mL
  Serotype Ia Day 1 | 0.24 [0.19 to 0.3] | 0.25 [0.2 to 0.32] | 0.38 [0.3 to 0.48]
  Serotype Ia Day 15 | 2.62 [1.64 to 4.17] | 2.95 [1.86 to 4.69] | 5.61 [3.56 to 8.84]
  Serotype Ia Day 31 | 2.68 [1.75 to 4.1] | 3.26 [2.14 to 4.98] | 6.63 [4.37 to 10]
  Serotype Ia At delivery | 2.22 [1.5 to 3.29] | 2.69 [1.82 to 3.98] | 4.49 [3.06 to 6.6]
  Serotype Ib Day 1 | 0.51 [0.38 to 0.7] | 0.36 [0.27 to 0.48] | 0.4 [0.31 to 0.51]
  Serotype Ib Day 15 | 2.93 [1.73 to 4.95] | 3.5 [2.17 to 5.65] | 6.07 [3.98 to 9.26]
  Serotype Ib Day 31 | 2.62 [1.62 to 4.24] | 3.68 [2.38 to 5.7] | 5.35 [3.63 to 7.87]
  Serotype Ib At delivery | 2.12 [1.36 to 3.31] | 3.04 [2.03 to 4.56] | 3.84 [2.69 to 5.5]
  Serotype III Day 1 | 0.12 [0.086 to 0.17] | 0.099 [0.072 to 0.14] | 0.14 [0.1 to 0.18]
  Serotype III Day 15 | 1.24 [0.79 to 1.95] | 1.52 [0.97 to 2.36] | 5.9 [3.99 to 8.72]
  Serotype III Day 31 | 1.51 [0.97 to 2.35] | 1.31 [0.85 to 2.02] | 5.35 [3.66 to 7.83]
  Serotype III At delivery | 1.25 [0.81 to 1.94] | 1.07 [0.7 to 1.65] | 3.8 [2.61 to 5.55]

3. Secondary Outcome: Percentages of Maternal Subjects With The Enzyme-linked Immunosorbent Assay (ELISA) Antibody Levels for GBS Serotypes Ia, Ib and III Above a Specific Threshold at Delivery
Description: Immunogenicity was measured in terms of the percentages of maternal subjects with ELISA Antibody Levels for GBS Serotypes Ia, Ib and III Above a Specific Threshold after receiving one dose of GBS Trivalent Vaccine.Threshold values of 0.1, 0.2, 0.5, 1, 2, 3, 5, and 8 μg/mL were used for serum concentrations for maternal subjects.
Time Frame: Day of Delivery
Population: FAS (Maternal Subjects)
Measure: Number; unit: Percentage of maternal subjects
Arm/Group | HIVposCD4LOW_Maternal | HIVposCD4HIGH_Maternal | HIVneg_Maternal
Number analyzed (Participants) | 83 | 82 | 83
Percentage of maternal subjects
  ≥ 0.2 µg/mL(Serotype Ia) | 100 | 99 | 100
  ≥ 0.5 µg/mL(Serotype Ia) | 67 | 71 | 82
  ≥ 1 µg/mL(Serotype Ia) | 55 | 59 | 71
  ≥ 2 µg/mL(Serotype Ia) | 51 | 49 | 60
  ≥ 3 µg/mL(Serotype Ia) | 40 | 46 | 54
  ≥ 5 µg/mL(Serotype Ia) | 30 | 41 | 53
  ≥ 8 µg/mL(Serotype Ia) | 22 | 30 | 47
  ≥ 0.1 µg/mL(Serotype Ib) | 89 | 98 | 98
  ≥ 0.2 µg/mL(Serotype Ib) | 88 | 98 | 98
  ≥ 0.5 µg/mL(Serotype Ib) | 83 | 84 | 90
  ≥ 1 µg/mL(Serotype Ib) | 65 | 63 | 69
  ≥ 2 µg/mL(Serotype Ib) | 40 | 41 | 47
  ≥ 3 µg/mL(Serotype Ib) | 28 | 35 | 40
  ≥ 5 µg/mL(Serotype Ib) | 20 | 26 | 28
  ≥ 8 µg/mL(Serotype Ib) | 13 | 17 | 24
  ≥ 0.1 µg/mL(Serotype III) | 96 | 80 | 95
  ≥ 0.2 µg/mL(Serotype III) | 82 | 76 | 89
  ≥ 0.5 µg/mL(Serotype III) | 63 | 51 | 86
  ≥ 1 µg/mL(Serotype III) | 47 | 41 | 73
  ≥ 2 µg/mL(Serotype III) | 36 | 24 | 64
  ≥ 3 µg/mL(Serotype III) | 29 | 18 | 54
  ≥ 5 µg/mL(Serotype III) | 18 | 13 | 49
  ≥ 8 µg/mL(Serotype III) | 17 | 12 | 40

4. Secondary Outcome: Percentages of Subjects With Solicited Local Adverse Events (AEs)
Description: Safety was assessed in terms of the number of subjects with solicited local AEs after receiving one dose of the GBS Trivalent Vaccine
Time Frame: From 6 Hours to Day 7 After Each Vaccination, for up to 24 weeks
Population: Safety Set (Solicited AEs, Maternal Subjects)
Measure: Number; unit: percentage of Subjects
Arm/Group | HIVposCD4LOW_Maternal | HIVposCD4HIGH_Maternal | HIVneg_Maternal
Number analyzed (Participants) | 88 | 88 | 90
percentage of Subjects
  Ecchymosis(87, 88, 90) | 0 | 0 | 1
  Erythema(87, 88, 89) | 0 | 1 | 1
  Induration(87, 88, 90) | 0 | 1 | 0
  Swelling(87, 88, 90) | 0 | 0 | 2
  Pain(87, 88, 90) | 18 | 30 | 39

5. Secondary Outcome: Percentages of Subjects With Solicited Systemic AEs
Description: Safety was assessed in terms of the number of subjects with solicited systemic AEs after receiving one dose of the GBS Trivalent Vaccine
Time Frame: From 6 Hours to Day 7 After Each Vaccination, for up to 24 weeks
Population: Safety Set (Solicited AEs, Maternal Subjects)
Measure: Number; unit: percentages of Subjects
Arm/Group | HIVposCD4LOW_Maternal | HIVposCD4HIGH_Maternal | HIVneg_Maternal
Number analyzed (Participants) | 88 | 88 | 90
percentages of Subjects
  Chills(87,88,90) | 9 | 14 | 22
  Nausea(87,88,89) | 13 | 17 | 22
  Malaise(87,88,90) | 10 | 19 | 23
  Myalgia(87,88,90) | 8 | 17 | 23
  Arthralgia(87,88,90) | 13 | 23 | 29
  Headache(87,88,90) | 24 | 32 | 43
  Fatigue(87,88,90) | 24 | 31 | 47
  Rash(87,88,90) | 3 | 1 | 1
  Fever ( ≥ 38°C)(87, 88, 90) | 3 | 0 | 0
  Temperature(<38°C)(87, 88,90) | 97 | 100 | 100
  Temperature(38-38.4°C)(87, 88,90) | 1 | 0 | 0
  Temperature(38.5-38.9°C)(87, 88,90) | 1 | 0 | 0
  Temperature(39-39.4°C)(87, 88,90) | 0 | 0 | 0
  Temperature(39.5-39.9°C)(87, 88,90) | 1 | 0 | 0
  Temperature(≥ 40°C)(87, 88,90) | 0 | 0 | 0
  Analgesic antipyr. meds(Other indicators) | 7 | 10 | 9
  Stayed home(Other indicators) | 3 | 5 | 9

6. Secondary Outcome: Percentages of Subjects Who Experienced Unsolicited Adverse Events
Description: Safety was assessed in terms of the number of subjects who experienced Unsolicited Adverse Events after receiving one dose of the GBS Trivalent Vaccine
Time Frame: Day 1 to Study Termination, for up to 24 weeks
Population: Safety Set (Unsolicited AEs, Maternal Subjects)
Measure: Number; unit: percentages of subjects
Arm/Group | HIVposCD4LOW_Maternal | HIVposCD4HIGH_Maternal | HIVneg_Maternal
Number analyzed (Participants) | 90 | 89 | 90
percentages of subjects
  Any AE | 74 | 76 | 78
  Possibly related AE | 7 | 13 | 23
  SAE | 28 | 31 | 32
  Possibly related SAE | 0 | 0 | 0
  AE leading to withdrawal from study | 0 | 1 | 0
  Medically attended AEs | 47 | 49 | 54
  Death | 0 | 1 | 0

7. Secondary Outcome: Percentages of Infants Who Experienced Unsolicited Adverse Events
Description: Safety in Infants was assessed in terms of the number of subjects who experienced Unsolicited Adverse Events since birth to study termination
Time Frame: Birth to Study Termination, for up to 24 weeks
Population: Safety Set (Unsolicited AEs, Infants)
Measure: Number; unit: percentages of Infant subjects
Arm/Group | HIVposCD4LOW (Infants) | HIVposCD4HIGH (Infants) | HIVneg (Infants)
Number analyzed (Participants) | 91 | 88 | 87
percentages of Infant subjects
  Any AE | 41 | 49 | 43
  Possibly related AE | 0 | 2 | 1
  SAE | 19 | 18 | 18
  Possibly related SAE | 0 | 0 | 0
  AE leading to withdrawal from study | 4 | 2 | 2
  Medically attended AEs | 23 | 33 | 24
  Death | 4 | 2 | 2

8. Primary Outcome: Geometric Mean Antibody Transfer Ratio Between Infant Antibody Level (μg/mL) and Maternal Antibody Level (μg/mL), for GBS Serotypes Ia, Ib and III at Delivery/Birth.
Description: The Geometric mean transfer ratio of GBS-specific Ab against serotypes Ia, Ib and III at delivery is calculated as the geometric mean of the pairwise ratios between the antibody concentrations from infant at birth and to maternal serum concentration at delivery.
Time Frame: Day of delivery/birth
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Groups:
- HIVposCD4LOW: Maternal Subjects:HIV-antibody positive maternal subjects at 24 to 35 weeks gestation with CD4+ count ≤350 cells/µL but > 50 cells/µL received one dose of 5 μg of each of the 3 glycoconjugates present in the GBS Trivalent Vaccine Infants:Infants born to HIV-antibody positive maternal subjects with CD4+ count ≤350 cells/µL but > 50 cells/µL
- HIVposCD4HIGH: Maternal Subjects:HIV-antibody positive maternal subjects at 24 to 35 weeks gestation with CD4+ count >350 cells/µL received one dose of 5 μg of each of the 3 glycoconjugates present in the GBS Trivalent Vaccine Infants:Infants born to HIV-antibody positive maternal subjects with CD4+ count >350 cells/µL
- HIVneg: Maternal subjects: HIV-antibody negative maternal subjects at 24 to 35 weeks gestation received one dose of 5 μg of each of the 3 glycoconjugates present in the GBS Trivalent Vaccine.
  Infants: Infants born to HIV-antibody negative maternal subjects
Arm/Group | HIVposCD4LOW | HIVposCD4HIGH | HIVneg
Number analyzed (Participants) | 79 | 79 | 83
Ratios
  Serotype Ia | 0.58 [0.49 to 0.69] | 0.6 [0.51 to 0.72] | 0.72 [0.61 to 0.85]
  Serotype Ib (41,54,57) | 0.51 [0.38 to 0.69] | 0.64 [0.5 to 0.83] | 0.49 [0.38 to 0.63]
  Serotype III (53,44,66) | 0.6 [0.44 to 0.82] | 0.51 [0.36 to 0.72] | 0.56 [0.43 to 0.75]
Statistical Analysis 1: Comparison: HIVposCD4LOW vs HIVposCD4HIGH; Test type: Superiority or Other; Vaccine Group Ratios (Serotype Ia) = 0.96, 98.4% CI 2-sided [0.71 to 1.3]
Statistical Analysis 2: Comparison: HIVposCD4LOW vs HIVneg; Test type: Superiority or Other; Vaccine Group ratios (Serotype Ia) = 0.81, 98.4% CI 2-sided [0.6 to 1.09]
Statistical Analysis 3: Comparison: HIVposCD4HIGH vs HIVneg; Test type: Superiority or Other; Vaccine Group ratios (Serotype Ia) = 0.84, 98.4% CI 2-sided [0.63 to 1.14]
Statistical Analysis 4: Comparison: HIVposCD4LOW vs HIVposCD4HIGH; Test type: Superiority or Other; Vaccine Group ratios (Serotype Ib) = 0.8, 98.4% CI 2-sided [0.49 to 1.29]
Statistical Analysis 5: Comparison: HIVposCD4LOW vs HIVneg; Test type: Superiority or Other; Vaccine Group ratios (Serotype Ib) = 1.05, 98.4% CI 2-sided [0.65 to 1.69]
Statistical Analysis 6: Comparison: HIVposCD4HIGH vs HIVneg; Test type: Superiority or Other; Vaccine Group ratios (Serotype Ib) = 1.32, 98.4% CI 2-sided [0.85 to 2.06]
Statistical Analysis 7: Comparison: HIVposCD4LOW vs HIVposCD4HIGH; Test type: Superiority or Other; Vaccine Group ratios (Serotype III) = 1.17, 98.4% CI 2-sided [0.66 to 2.07]
Statistical Analysis 8: Comparison: HIVposCD4LOW vs HIVneg; Test type: Superiority or Other; Vaccine Group ratios (Serotype III) = 1.06, 98.4% CI 2-sided [0.63 to 1.78]
Statistical Analysis 9: Comparison: HIVposCD4HIGH vs HIVneg; Test type: Superiority or Other; Vaccine Group ratios (Serotype III) = 0.91, 98.4% CI 2-sided [0.52 to 1.58]

ADVERSE EVENTS:
Time Frame: Throughout the study period, for up to 24 weeks
Description: All AEs or SAEs occurring from previous visit, relevant medical history, any new or continuing concomitant medications were recorded at the next visit. All AEs were collected until day 31 following vaccination and all AEs requiring a physician's visit from day 31 until the end of study. All SAEs were monitored throughout the entire study period.
Groups:
- HIVposCD4LOW (Infants): Infants born to HIV-antibody positive maternal subjects with CD4+ count ≤350 cells/μL but > 50 cells/μL
- HIVposCD4HIGH (Infants): Infants born to HIV-antibody positive maternal subjects with CD4+ count >350 cells/μL .
- Total (Infants): Total number of Infants participated in the study
- HIVposCD4LOW_Maternal Subjects: HIV-antibody positive maternal subjects at 24 to 35 weeks gestation with CD4+ count ≤350 cells/μL but > 50 cells/μL received one dose of 5 μg of each of the 3 glycoconjugates present in the GBS Trivalent vaccine.
- HIVposCD4HIGH_Maternal Subjects: HIV-antibody positive maternal subjects at 24 to 35 weeks gestation with CD4+ count >350 cells/μL received one dose of 5 μg of each of the 3 glycoconjugates present in the GBS Trivalent vaccine.
- HIVneg_Maternal Subjects: HIV-antibody negative maternal subjects at 24 to 35 weeks gestation received one dose of 5 μg of each of the 3 glycoconjugates present in the GBS Trivalent vaccine.
- Total Maternal Subjects: Total number of Maternal subjects participated in the study
Arm/Group | HIVposCD4LOW (Infants) | HIVposCD4HIGH (Infants) | HIVneg (Infants) | Total (Infants) | HIVposCD4LOW_Maternal Subjects | HIVposCD4HIGH_Maternal Subjects | HIVneg_Maternal Subjects | Total Maternal Subjects
Serious Adverse Events (participants affected / at risk) | 17/91 | 16/88 | 16/87 | 49/266 | 25/90 | 28/89 | 29/90 | 82/269
Other Adverse Events (participants affected / at risk) | 13/91 | 11/88 | 7/87 | 31/266 | 55/90 | 68/89 | 71/90 | 194/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIVposCD4LOW (Infants) (N=91) | HIVposCD4HIGH (Infants) (N=88) | HIVneg (Infants) (N=87) | Total (Infants) (N=266) | HIVposCD4LOW_Maternal Subjects (N=90) | HIVposCD4HIGH_Maternal Subjects (N=89) | HIVneg_Maternal Subjects (N=90) | Total Maternal Subjects (N=269)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 1
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
HAEMORRHAGIC DISEASE OF NEWBORN (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
CARDIAC ARREST (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
CARDIAC DISORDER (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CHROMOSOMAL DELETION (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CONGENITAL PNEUMONIA (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
PATENT DUCTUS ARTERIOSUS (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
TALIPES (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
TRISOMY 21 (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
FEELING JITTERY (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
AMNIOTIC CAVITY INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
BREAST ABSCESS (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
ENDOMETRITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
MALARIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
MENINGITIS (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 2 | 0 | 1 | 3 | 0 | 0 | 0 | 0
POST PROCEDURAL SEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
SEPSIS (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SEPSIS NEONATAL (Infections and infestations) | 3 | 5 | 3 | 11 | 0 | 0 | 0 | 0
SYPHILIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
PERINEAL INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
UTERINE RUPTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
BLOOD PRESSURE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
HAEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
CONVULSION (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
EPILEPSY (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
HYPOXIC-ISCHAEMIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0 | 3 | 4 | 0 | 0 | 0 | 0
PARTIAL SEIZURES (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
VIITH NERVE PARALYSIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
BREECH PRESENTATION (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
CAPUT SUCCEDANEUM (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
CEPHALO-PELVIC DISPROPORTION (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 3 | 0 | 9 | 12
CERVIX DYSTOCIA (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
ECLAMPSIA (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
FAILED INDUCTION OF LABOUR (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
FALSE LABOUR (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
FOETAL DISTRESS SYNDROME (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 2 | 6 | 2 | 1 | 9
GESTATIONAL DIABETES (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
GESTATIONAL HYPERTENSION (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 4
HAEMORRHAGE IN PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 6
HYPEREMESIS GRAVIDARUM (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
JAUNDICE NEONATAL (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 2 | 4 | 0 | 0 | 0 | 0
LOW BIRTH WEIGHT BABY (Pregnancy, puerperium and perinatal conditions) | 2 | 2 | 1 | 5 | 0 | 0 | 0 | 0
POSTPARTUM HAEMORRHAGE (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
PRE-ECLAMPSIA (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3
PREMATURE BABY (Pregnancy, puerperium and perinatal conditions) | 5 | 3 | 3 | 11 | 0 | 0 | 0 | 0
PREMATURE DELIVERY (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 6
PREMATURE LABOUR (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 7
PRETERM PREMATURE RUPTURE OF MEMBRANES (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 3 | 7 | 2 | 12
PROLONGED LABOUR (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 3 | 5 | 5 | 13
PROLONGED PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
PROLONGED RUPTURE OF MEMBRANES (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 4
RETAINED PLACENTA OR MEMBRANES (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
RETAINED PRODUCTS OF CONCEPTION (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
STILLBIRTH (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
THREATENED LABOUR (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3
TRANSVERSE PRESENTATION (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
UTERINE CERVIX STENOSIS (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
NEONATAL ASPHYXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 5 | 0 | 0 | 0 | 0
NEONATAL ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 4 | 0 | 0 | 0 | 0
NEONATAL RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 7 | 0 | 0 | 0 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
TRANSIENT TACHYPNOEA OF THE NEWBORN (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 0
MELANOSIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CAESAREAN SECTION (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 6
HAEMATOMA (Vascular disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
SHOCK (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
SHOCK HAEMORRHAGIC (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
SUBGALEAL HAEMATOMA (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HIVposCD4LOW (Infants) (N=91) | HIVposCD4HIGH (Infants) (N=88) | HIVneg (Infants) (N=87) | Total (Infants) (N=266) | HIVposCD4LOW_Maternal Subjects (N=90) | HIVposCD4HIGH_Maternal Subjects (N=89) | HIVneg_Maternal Subjects (N=90) | Total Maternal Subjects (N=269)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 3 | 5 | 10
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 7 | 8
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 12 | 16 | 22 | 50
CHILLS (General disorders) | 0 | 0 | 0 | 0 | 8 | 12 | 20 | 40
FATIGUE (General disorders) | 0 | 0 | 0 | 0 | 21 | 27 | 42 | 90
INJECTION SITE PAIN (General disorders) | 0 | 0 | 0 | 0 | 16 | 27 | 36 | 79
MALAISE (General disorders) | 0 | 0 | 0 | 0 | 9 | 18 | 21 | 48
PAIN (General disorders) | 0 | 0 | 0 | 0 | 3 | 3 | 5 | 11
CONJUNCTIVITIS (Infections and infestations) | 7 | 3 | 2 | 12 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 | 6 | 3 | 19 | 9 | 9 | 1 | 19
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 6 | 5 | 1 | 12
PERINEAL INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 17 | 24 | 21 | 62
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 11 | 20 | 26 | 57
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 7 | 15 | 21 | 43
HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 23 | 32 | 41 | 96
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 4 | 3 | 2 | 5 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.